CLINICAL TRIAL: NCT06394011
Title: A Single-center, Single-arm, Prospective Clinical Study on the Efficacy and Safety of Venetoclax and Azacitidine Combined With HAAG in the Induction Treatment of Intermediate and High-risk Acute Myeloid Leukemia
Brief Title: Study of VA Combined With HAAG Regimen in Newly Diagnosed Intermediate and High-risk AML Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VA+HAAG
Record Dates: First submitted 2024-04-27; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-01

CONDITIONS: Intermediate Risk Acute Myeloid Leukemia; High Risk Acute Myeloid Leukemia
MeSH Terms: interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VA combined with HAAG (Experimental): This cohort will determine the safety and efficacy of venetoclax, azacitidine combined with HAAG regimen in newly diagnosed intermediate and high-risk AML patients.
  Interventions: Drug: venetoclax, azacitidine and HAAG regimen

INTERVENTIONS:
Drug: venetoclax, azacitidine and HAAG regimen — Venetoclax:100mg, qd, d1;200mg, qd, d2;400 mg, qd, d3~10, per os; Azacitidine:75mg/m2/d, d1~7, subcutaneous injection; Homoharringtonine:1mg/d, d4~10, intravenous infusion; Aclarubicin:10mg/d, d4~7, intravenous infusion; Cytarabine:10mg/m2,q12h,d4~10, subcutaneous injection; Granulocyte colony-stimulating factor (G-CSF): 50-300μg/d (when WBC counts are less than 20×10^9/L ),subcutaneous injection;

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of VA combined with HAAG in the induction treatment of newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective clinical study in newly diagnosed intermediate and high-risk AML patients. The patients will receive venetoclax, azacitidine combined with HAAG regimen in the induction treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed intermediate and high-risk AML according to the WHO (2022) classification of acute myeloid leukemia (non-APL).
2. Age 18-65.
3. ECOG score: 0-2.
4. No history of previous chemotherapy or target therapy.
5. Serum total bilirubin <= 2 times the upper limit of normal (ULN), alanine aminotransferase (ALT) <= 1.5 times ULN, aspartate aminotransferase (AST) <=1.5 times ULN;
6. Creatinine clearance rate >=30 mL/min;
7. Serum lipase <= 1.5 times ULN, amylase <= 1.5 times ULN;
8. Capable to understand and willing to participate in this study, signed the informed consent form.

Exclusion Criteria:

1. AML transformed with chronic myelogenous leukemia.
2. Acute promyelocytic leukemia (type M3).
3. Patients with a second malignancy requiring treatment.
4. Patients with uncontrolled active infection.
5. Patients with left ventricular ejection fraction < 0.5 by echocardiography or grade III/IV cardiovascular dysfunction according to the New York Heart Association Classification.
6. Patients with hepatic and renal inadequacy: total serum bilirubin >=2.0 mg/dl, AST >=3 times ULN, serum creatinine clearance (Ccr) <50 ml / min.
7. Patients with arterial oxygen saturation (SpO 2) was <95%.
8. Patients with HIV infection.
9. Patients with active hepatitis B or hepatitis C infection.
10. Patients with other commodities that the investigators considered not suitable for the enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite complete response rate (CRc; CR+CRi) | Day 28-35 of induction course
  CRc includes complete response CR and CRi; CR was defined as < 5% bone marrow blasts in an aspirate with spicules, no blasts with Auer rods or persistence of extramedullary disease, and independent of transfusions; CRi: was defined as<5% bone marrow blasts, either ANC<1×10^9/L or platelets<100×10^9/L, transfusion independence but with persistence of cytopenia.

SECONDARY OUTCOMES:
Partial remission (PR) | Day 28-35 of induction course
  PR was defined as decrease of at least 50% in the percentage of blasts to 5-25% in the bone marrow aspirate and the normalization of blood counts.
Number of adverse events | 2 years
  adverse events are evaluated with CTCAE V5.0.
Relapse-free survival (RFS) | 3 years
  time from clinical CRc (CR and CRi) to the first relapse or death
Overall survival (OS) | 3 years
  time from the first day of treatment to death or lost to follow-up for any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowen Tang, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China